CLINICAL TRIAL: NCT04363437
Title: COlchicine in Moderate-severe Hospitalized Patients Before ARDS to Treat COVID-19 (the COMBAT-COVID-19 Pilot Study)
Brief Title: COlchicine in Moderate-severe Hospitalized Patients Before ARDS to Treat COVID-19
Acronym: COMBATCOVID19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped due to widespread corticosteroid use in 2020 for COVID infection, which confounds and likely supercedes the effect of colchicine.
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-04-12
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus Infection
Keywords: colchicine; anti-inflammatory
MeSH Terms: conditions — Coronavirus Infections | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchine (Active Comparator)
  Interventions: Drug: Colchicine
- Usual Care (Active Comparator)
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: Colchicine — People in the colchine group will be given a starting dose of 1.2 mg followed, by 0.6mg after 2 hours if they do not have significant gastrointestinal symptoms, on day 1. After that, they will take colchicine 0.6mg twice a day for 14 days or until discharged or release from the hospital.
  Arms: Colchine
Drug: Usual Care — COVID Patients in this arm will receive usual care COVID19 treatment and will not receive colchine.
  Arms: Usual Care

SUMMARY:
The most prevalent complication of COVID-19 infection is respiratory failure from severe acute respiratory syndrome (SARS), the leading cause of mortality. There is increasing indication that the decompensation in severe COVD-19 infection may be due to a cytokine storm syndrome. This hyperinflammatory syndrome results in a fulminant and fatal hypercytokinemia and multiorgan failure.

Approximately 15% of patients with COVID-19 infection are hospitalized and 20-30% of these hospitalized patients require ICU care and/or mechanical ventilation. Overall mortality in hospitalized patients is approximately 20-25%. There is significant interest in therapies that can be given upstream to reduce the rate of mechanical ventilation and thus mortality.

We hypothesize that treatment with colchicine in COVID-19 moderate-severe patients may decrease the risk of progression into ARDS requiring increased oxygen requirements, mechanical ventilation, and mortality.

DETAILED DESCRIPTION:
Prospective, completely randomized, open labeled, controlled study. Patients will be randomized into two groups (A and B). Patients of group A will be treated under what is considered current standard of care at Maimonides Medical Center while group B patients will receive colchicine in addition to standard of care.

Treatment arm

In addition to the local standard of care for COVID 19 patients, the patient will receive colchicine PO as such:

* Loading dose of 1.2 mg followed by 0.6mg after 2 hours if without significant gastrointestinal symptoms (day 1)
* The next day 0.6mg bid for 14 days or until discharge

Patients who are on HMG-Co A Reductase Inhibitors (atorvastatin, fluvastatin, pravastatin, simvastatin), fibrates, genfibrozil, amiodarone, dronedarone or digoxin should have the colchicine dosage reduced to a loading dose of 0.6mg followed by 0.3mg after two hours (day 1) followed by 0.3mg BID for 14 days or until discharge.

If patients have significant gastrointestinal symptoms after loading, the dosage may be reduced to 0.3mg BID for the rest of the 14 day course or until discharge. If gastrointestinal symptoms continue, the medication should then be discontinued. Patients who experience sensory motor neuropathy, or symptoms and laboratory findings consistent with rhabdomyolysis should prompt immediate discontinuation of the drug. If renal function deteriorates during the treatment course and CrCl <30ml/min, colchicine should also be discontinued.

Control arm Usual medical therapy (can include medications such as hydroxychloroquine, azithromycin)

Patients should NOT receive, Remdesivir, IL-6 inhibitors (Tociluzimab, Sarilumab), JAK inhibitors, IL-1 inhibitors, or other immunomodulators for COVID-19 before randomization. Since the primary clinical endpoint is progression of disease, if the patient requires beyond 8L nasal cannula, eg. high flow O2 or mechanical ventilation, the primary clinical endpoint is met and the above experimental medications will be permitted. To rephrase, the patient will be allowed, Remdesivir, IL-6 inhibitors and other immunomodulators if then deemed medically necessary by the treating physician.

ELIGIBILITY:
* Males and females >=18 years of age
* Willing and able to provide written informed consent prior to performing study procedures
* Currently hospitalized and requiring medical care for COVID-19
* Significant COVID-19 symptom, or judged by the treating provider to be at high risk of progression to severe COVID-19 infection
* Significant COVID-19 symptoms are defined by one or more of the following:

  1. Dyspnea
  2. Respiratory frequency ≥ 30/min
  3. Blood oxygen saturation ≤ 93%
* AND one or more of the following: (positive PCR test or positive antibodies) or (CT/Chest X-ray consistent with COVID19 infection) or (anosmia).

Exclusion Criteria:

* Requirement of oxygen supplementation >8L nasal cannula
* Pregnancy
* Known hypersensitivity to colchicine
* Patient currently in shock or with hemodynamic instability requiring pressors
* History of cirrhosis
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5X upper limit of normal (ULN)
* Patients with severe renal disease, CrCl <30ml/min
* Patients requiring invasive mechanical ventilation at screening or Clinical estimation that the patient will require mechanical respiratory support within 24 hours
* Patient is currently taking colchicine for other indications (gout or Familial Mediterranean Fever)
* Patient received Remdesivir, Sarilumab, Tociluzimab, Lopinavir/Ritonavir or other immunomodulator given for COVID-19 treatment (Note: Convalescent plasma infusion is not an exclusion)
* Patient is on (and cannot discontinue) a strong CYP3A4 inhibitor (eg clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, atazanavir), a moderate CYP3A4 inhbitor (eg diltiazem, verapamil, fluconazole, amprenavir, aprepitant, fosamprenavir) or a P-gp Inhibitor (eg cyclosporine, ranolazine)
* Patient is undergoing chemotherapy for cancer
* Patient is considered by the investigator, for any reason, to be unsuitable candidate for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-04-26 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Yang, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colchine | Usual Care
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchine | Usual Care | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (18.1) | 67.1 (20.4) | 64.47 (19.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Requiring Supplemental Oxygen Beyond 8L Nasal Cannula
Time Frame: through study completion, estimated 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Colchine | Usual Care
Number analyzed (Participants) | 10 | 11
Participants | 1 | 1

2. Secondary Outcome: Percentage of Patients Who Will Require Mechanical Ventillation
Time Frame: through study completion, estimated 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Colchine | Usual Care
Number analyzed (Participants) | 10 | 11
Participants | 1 | 0

3. Secondary Outcome: Mortality
Time Frame: through study completion, estimated 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Colchine | Usual Care
Number analyzed (Participants) | 10 | 11
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Colchine | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04363437/Prot_SAP_002.pdf